CLINICAL TRIAL: NCT00266253
Title: A Randomized Double-blind Study to Determine the Effect of GK Activator (2) on Efficacy (HbA1c), Safety, Tolerability and Pharmacokinetics in Patients With Type 2 Diabetes Mellitus Treated With a Stable Dose of Metformin.
Brief Title: A Study of GK Activator (2) in Patients With Type 2 Diabetes Mellitus Treated With a Stable Dose of Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM18249
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Metformin
- 2 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Metformin
- 3 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Metformin
- 4 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Metformin
- 5 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Metformin
- 6 (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: GK Activator (2) — Escalating doses, po bid or qd for 12 weeks.
  Arms: 1; 2; 3; 4; 5
Drug: Metformin — As prescribed, for 12 weeks

SUMMARY:
This study will evaluate the efficacy, safety, tolerability, and pharmacokinetics of GK Activator (2) in combination with metformin, compared to that of placebo (metformin monotherapy), in patients with type 2 diabetes mellitus. Patients will continue on their stable dose of metformin and will be randomized to receive either GK Activator (2) or placebo. The anticipated time on study treatment is less than 3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 30-75 years of age;
* type 2 diabetes mellitus;
* individual maximal tolerated daily dose of metformin monotherapy for >=3 months prior to screening.

Exclusion Criteria:

* type 1 diabetes mellitus;
* any oral anti-hyperglycemic medication, other than metformin monotherapy, during last 3 months

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2005-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
HbA1c mean change from baseline compared with placebo. | Week 12

SECONDARY OUTCOMES:
Additional parameters of glycemic and lipid control. | Week 12
AEs, laboratory parameters. | Throughout study
Pharmacokinetic and exposure-response relationship | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (47):
- United States (18):
  - Phoenix, Arizona
  - Chula Vista, California
  - Los Angeles, California
  - Kissimmee, Florida
  - Tampa, Florida
  - Lawrenceville, Georgia
  - Arkansas City, Kansas
  - Benzonia, Michigan
  - Springfield, Missouri
  - Butte, Montana
  - Kettering, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Morrisville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Bellevue, Washington
  - Federal Way, Washington
- Australia (3):
  - Adelaide
  - Heidelberg
  - Sydney
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Germany (10):
  - Bammental
  - Berlin
  - Essen
  - Giessen
  - Görlitz
  - Hamburg
  - Künzing
  - Mannheim
  - Nuremberg
  - Tann
- Spain (4):
  - Alzira
  - Bacarot Alicant
  - Barakaldo
  - Barcelona
- United Kingdom (7):
  - Dundee
  - Frome
  - Glasgow
  - Liverpool
  - Motherwell
  - Northwood
  - Plymouth